CLINICAL TRIAL: NCT03646123
Title: Multiple Part Clinical Trial of Brentuximab Vedotin in Classical Hodgkin Lymphoma Subjects
Brief Title: Clinical Trial of Brentuximab Vedotin in Classical Hodgkin Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was prematurely discontinued as the sponsor believes the data collected is enough to show the safety and efficacy of the combinations studied in all cohorts. The decision was not based on any safety and/or efficacy concerns.
Sponsor: Seagen Inc. (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGN35-027
Record Dates: First submitted 2018-08-22; First posted 2018-08-24 (Actual); Results first posted 2023-12-21 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Hodgkin Lymphoma
Keywords: Brentuximab vedotin; Doxorubicin; Vinblastine; Dacarbazine; Nivolumab; Seattle Genetics
MeSH Terms: conditions — Hodgkin Disease | interventions — Brentuximab Vedotin; Doxorubicin; Vinblastine; Dacarbazine; Granulocyte Colony-Stimulating Factor; Filgrastim; pegfilgrastim; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: A+AVD (Experimental): Brentuximab vedotin (A) plus doxorubicin (+A), vinblastine (V), and dacarbazine (D) administered by intravenous (IV) infusion in participants with advanced stage classical Hodgkin lymphoma (cHL) during each treatment cycle.
  Interventions: Drug: brentuximab vedotin; Drug: doxorubicin; Drug: vinblastine; Drug: dacarbazine; Drug: G-CSF
- Part B: AN+AD (Experimental): Brentuximab vedotin (A) plus nivolumab (N), doxorubicin (+A), and dacarbazine (D) administered separately by IV infusion in participants with Stage II bulky mediastinal disease and Stage III or IV cHL during each treatment cycle.
  Interventions: Drug: brentuximab vedotin; Drug: doxorubicin; Drug: dacarbazine; Drug: nivolumab
- Part C: AN+AD (Experimental): Brentuximab vedotin (A) plus nivolumab (N), doxorubicin (+A), and dacarbazine (D) administered separately by IV infusion in participants with Stage I or II cHL with non-bulky mediastinal disease during each treatment cycle.
  Interventions: Drug: brentuximab vedotin; Drug: doxorubicin; Drug: dacarbazine; Drug: nivolumab

INTERVENTIONS:
Drug: brentuximab vedotin — 1.2 mg/kg by IV infusion
  Other Names: Adcetris; SGN-35
Drug: doxorubicin — 25 mg/m^2 by IV infusion
Drug: vinblastine — 6 mg/m^2 by IV infusion
  Arms: Part A: A+AVD
Drug: dacarbazine — 375 mg/m^2 by IV infusion
Drug: G-CSF — Granulocyte colony stimulating factor (G-CSF) primary prophylaxis administered 24-36 hours after each dose of A+AVD
  Other Names: filgrastim; pegfilgrastim
  Arms: Part A: A+AVD
Drug: nivolumab — 240 mg by IV infusion
  Other Names: Opdivo
  Arms: Part B: AN+AD; Part C: AN+AD

SUMMARY:
This trial will study two treatment combinations for classical Hodgkin lymphoma (cHL). This trial will find out if these two treatment combinations work to treat cHL. It will also find out what side effects occur. A side effect is anything the drug does besides treating cancer. This study will have three parts (Parts A, B, and C).

The drugs used in Part A are a combination of targeted anticancer drug (brentuximab vedotin) and three chemotherapy drugs (doxorubicin, vinblastine, and dacarbazine). These four drugs are called "A+AVD." Participants will be treated with granulocyte colony stimulating factor (G-CSF) following every dose of A+AVD for 6 cycles of treatment (12 doses).

Part A will look at whether the A+AVD drug combination reduces the number of participants who experience the side effect of febrile neutropenia. Febrile neutropenia is a very low white blood cell count and a fever, which can be life threatening.

Parts B and C will use drug combination of brentuximab vedotin, plus nivolumab, doxorubicin, and dacarbazine. These four drugs are called "AN+AD." Parts B and C will study how well the drugs work to treat cHL and what side effects they cause.

DETAILED DESCRIPTION:
This study will have three parts.

Part A of the study is designed to evaluate the incidence of febrile neutropenia, efficacy, and dose intensity in participants with advanced stage classical Hodgkin lymphoma (cHL) receiving granulocyte colony stimulating factor primary prophylaxis (G-PP) administration during treatment with frontline A+AVD. In Part A, participants will be treated with granulocyte colony stimulating factor (G-CSF) following every dose of A+AVD for 6 cycles of treatment. Participants will be treated using institutional standard of care practices for the majority of treatment decisions.

Part B is designed to evaluate the combination of brentuximab vedotin, nivolumab, doxorubicin, and dacarbazine (AN+AD) as frontline treatment in participants with advanced cHL. In Part B, participants will be given AN+AD combination for 6 cycles of treatment. This part of the trial will look at whether this combination of drugs is effective and tolerable in participants with Stage II with bulky mediastinal disease and Stage III or IV cHL.

Part C is designed to evaluate AN+AD as frontline treatment in participants with early stage cHL. In Part C, participants will be given AN+AD combination for 4 cycles of treatment. This part of the trial will look at whether this combination of drugs is effective and tolerable in participants with Stage I or II cHL with non-bulky mediastinal disease.

ELIGIBILITY:
Inclusion Criteria

* Treatment-naïve, classic Hodgkin lymphoma (cHL) participants

  * Participants enrolling in Part A of the study must have Ann Arbor Stage III or IV disease
  * Participants enrolling in Part B of the study must have Ann Arbor Stage I or II cH: with bulky mediastinal disease, or Stage III or IV
  * Participants enrolling in Part C of the study must have Ann Arbor Stage I or II cHL without bulky disease
* Histologically confirmed cHL according to the current World Health Organization (WHO) Classification
* Bidimensional measurable disease as documented by PET/CT or CT imaging
* Age 12 years or older in the United States. For regions outside of the US, participants must 18 years or older.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2

Exclusion Criteria

* Nodular lymphocyte predominant HL
* History of another malignancy within 3 years of the first dose of study drug or any evidence of residual disease from a previously diagnosed malignancy. Exceptions are malignancies with a negligible risk or metastasis or death. Participants with nonmelanoma skin cancer, localized prostate cancer, or carcinoma in situ of any type are not excluded if they have undergone complete resection
* Prior immunosuppressive chemotherapy, therapeutic radiation, or any immunotherapy within 4 weeks of the first study drug dose
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
* Active cerebral/meningeal disease related to the underlying malignancy
* Any active Grade 3 or higher viral, bacterial, or fungal infection within two weeks of the first dose of study drug (Grade 3 defined by the National Cancer Institute's Common Terminology Criteria for Adverse Events, NCI CTCAE Version 4.03)
* Current therapy with other systemic anti-neoplastic or investigational agents
* Planned consolidative radiotherapy (Parts B and C only)
* Active interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity (Parts B and C only)
* Grade 3 or higher pulmonary disease unrelated to underlying malignancy
* Documented history of idiopathic interstitial pneumonia or diffusing capacity of the lung for carbon monoxide <50% predicted
* History of a cerebral vascular event within 6 months of first dose of study drug
* Child-Pugh B or C hepatic impairment
* Grade 2 or higher peripheral sensory or motor neuropathy
* Participants with acute or chronic graft-versus-host-disease (GvHD) or receiving immunosuppressive therapy as treatment or as prophylaxis against GvHD
* Previous treatment with brentuximab vedotin
* Participants who are pregnant or breastfeeding
* Other serious condition that would impair the participant's ability to receive or tolerate the planned treatment and follow-up

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2024-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Seagen Inc.
Locations (76):
- United States (55):
  - Los Angeles Cancer Network / Compassionate Care Research Group, Fountain Valley, California
  - Rocky Mountain Cancer Centers - Aurora, Aurora, Colorado
  - University of Colorado Health Memorial Hospital, Colorado Springs, Colorado
  - Cancer Centers of Colorado - Denver, Denver, Colorado
  - Poudre Valley Health System (PVHS), Fort Collins, Colorado
  - SCL Health - St. Mary's Hospital & Medical Center, Grand Junction, Colorado
  - Miami Cancer Institute at Baptist Health, Inc., Miami, Florida
  - Florida Cancer Specialists - North Region, St. Petersburg, Florida
  - Cardinal Bernardin Cancer Center / Loyola University Medical Center, Maywood, Illinois
  - Illinois Cancer Specialists, Niles, Illinois
  - Illinois Cancer Care, Peoria, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Karmanos Cancer Institute / Wayne State University, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Minnesota Oncology Hematology P.A., Edina, Minnesota
  - Washington University in St Louis, St Louis, Missouri
  - New Jersey Hematology Oncology Associates, LLC, Brick, New Jersey
  - Regional Cancer Care Associates - Freehold, Freehold, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Regional Cancer Care Associates - Howell, Howell Township, New Jersey
  - Morristown Medical Center/ Carol G. Simon Cancer Center, Morristown, New Jersey
  - Regional Cancer Care Associates - Mount Holly, Mount Holly, New Jersey
  - Regional Cancer Care Associates - Central Jersey, Somerville, New Jersey
  - Regional Cancer Care Associates - Sparta, Sparta, New Jersey
  - New York Oncology Hematology, P.C., Albany, New York
  - CareMount Medical Group, Mount Kisco, New York
  - Mount Sinai Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Clinical Research Alliance - Abraham Mittelman, MD, LLC, Purchase, New York
  - Clinical Research Alliance - Morton Coleman, MD, Westbury, New York
  - Wake Forest Baptist Medical Center / Wake Forest University, Winston-Salem, North Carolina
  - Oncology Hematology Care, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, The, Cleveland, Ohio
  - Toledo Clinic Cancer Center, Toledo, Ohio
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Medical University of South Carolina/Hollings Cancer Center, Charleston, South Carolina
  - University of Tennessee, Knoxville, Tennessee
  - Tennessee Oncology-Nashville/Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology - Austin Midtown, Austin, Texas
  - Texas Oncology - Medical City Dallas, Dallas, Texas
  - Texas Oncology - Flower Mound, Flower Mound, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Texas Oncology - Fort Worth 12th Avenue, Fort Worth, Texas
  - MD Anderson Cancer Center / University of Texas, Houston, Texas
  - Texas Oncology - San Antonio Medical Center, San Antonio, Texas
  - Texas Oncology - Northeast Texas, Tyler, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Oncology and Hematology Assoc of SW VA DBA Blue Ridge Cancer Care, Salem, Virginia
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Vista Oncology Inc PS, Olympia, Washington
  - Seattle Cancer Care Alliance / University of Washington, Seattle, Washington
- Australia (4):
  - Royal Adelaide Hospital, Adelaide, Other
  - Ballarat Regional Integrated Cancer Care, Ballarat, Other
  - Monash Medical Centre, Clayton, Other
  - Epworth Healthcare, Victoria, Other
- Czechia (2):
  - Fakultni nemocnice Hradec Kralove-oddeleni klinicke hematologie, Hradec Králové, Other
  - Fakultni Nemocnice Kralovske Vinohrady, Prague, Other
- Italy (4):
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia, Other
  - IRCSS Policlinico San Matteo, Pavia, Other
  - Azienda Ospedaliera Universitaria Senese, Siena, Other
  - Azienda Ospedaliera Citta della Salute e della Scienza di Torino, Torino, Other
- Pratia MCM Krakow, Krakow, Other, Poland
- Spain (10):
  - Hospital del Mar, Barcelona, Other
  - Hospital Universitari Vall d'Hebron, Barcelona, Other
  - Institut Catala d'Oncologia - Hospital Duran i Reynals (ICO L'Hospitalet), Barcelona, Other
  - Hospital Universitario de Girona Doctor Josep Trueta, Girona, Other
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid, Other
  - Hospital Universitario 12 de Octubre, Madrid, Other
  - Hospital Puerta de Hierro Majadahonda, Majadahonda, Other
  - Hospital Universitario Central de Asturias, Oviedo, Other
  - Hospital Clinico Universitario de Salamanca, Salamanca, Other
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia, Other

REFERENCES:
- [Derived] Abramson JS, Straus DJ, Bartlett NL, Burke JM, Lynch RC, Domingo-Domenech E, Hess BT, Schuster SR, Linhares Y, Gandhi MD, Shah HR, Jurczak W, Re A, Hahn U, Prince HM, Guo W, Davis G, Ho L, Fanale M, Yasenchak CA, Lee HJJ. Brentuximab Vedotin and Nivolumab in Combination With Chemotherapy for Nonbulky, Early-Stage Classical Hodgkin Lymphoma. Blood. 2025 Dec 29:blood.2025030190. doi: 10.1182/blood.2025030190. Online ahead of print. PMID 41460964
- [Derived] Lee HJ, Ramchandren R, Friedman J, Melear J, Flinn IW, Burke JM, Linhares Y, Gonzales P, Peterson M, Raval M, Chintapatla R, Feldman TA, Yimer H, Islas-Ohlmayer M, Patel A, Metheny L, Dean A, Rana V, Gandhi MD, Renshaw J, Ho L, Fanale MA, Guo W, Yasenchak CA. Brentuximab vedotin, nivolumab, doxorubicin, and dacarbazine for advanced-stage classical Hodgkin lymphoma. Blood. 2025 Jan 16;145(3):290-299. doi: 10.1182/blood.2024024681. PMID 39622165

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this study participant's treatment was completed before primary completion date (PCD), and no treatment was administered after PCD, participants were followed up.
Groups:
- Part A: A+AVD (brentuximab vedotin plus doxorubicin, vinblastine, and dacarbazine) in participants with advanced stage classical Hodgkin lymphoma (cHL).
- Part B: AN+AD (brentuximab vedotin and nivolumab plus doxorubicin and dacarbazine) in participants with Stage II bulky mediastinal disease and Stage III or IV cHL.
- Part C: AN+AD (brentuximab vedotin and nivolumab plus doxorubicin and dacarbazine) in participants with Stage I or II cHL with non-bulky mediastinal disease.
Period: Overall Study
Arm/Group | Part A | Part B | Part C
Started | 41 | 58 | 156
Treated | 40 | 57 | 154
Completed | 31 | 0 | 1
Not Completed | 10 | 58 | 155
Not completed — Withdrawal by Subject | 2 | 2 | 3
Not completed — Study termination by sponsor | 0 | 45 | 139
Not completed — Lost to Follow-up | 4 | 10 | 10
Not completed — Death | 2 | 1 | 1
Not completed — Other | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A | Part B | Part C | Total
Number analyzed (Participants) | 41 | 58 | 156 | 255
Age, Continuous [Median (Full Range); unit: years] | 28 [18 to 71] | 35 [19 to 78] | 31 [18 to 77] | 31 [18 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 27 | 86 | 129
  Male | 25 | 31 | 70 | 126
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 10 | 22 | 36
  Not Hispanic or Latino | 34 | 46 | 127 | 207
  Unknown or Not Reported | 3 | 2 | 7 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 1 | 1 | 6 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 2 | 1 | 9
  White | 31 | 50 | 131 | 212
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 3 | 4 | 17 | 24
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — 0=Normal activity; 1=Symptoms but ambulatory; 2=In bed <50% of the time; 3= In bed >50% of the time; 4=100% bedridden; 5=Dead
  Participants
    Grade 0 | 27 | 34 | 124 | 185
    Grade 1 | 13 | 23 | 28 | 64
    Grade 2 | 0 | 0 | 2 | 2
    Missing | 1 | 1 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Febrile Neutropenia (FN) Rate (Part A)
Description: The FN rate is defined as the number of participants who experience treatment-emergent FN.
Time Frame: 7.5 months
Population: For Part A, the full analysis set included all participants who received at least 1 dose of A+AVD (any of the study drugs in the regimen).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A
Number analyzed (Participants) | 40
Participants
  Any treatment-emergent FN | 5
  Treatment-related treatment-emergent FN | 5
  Grade 3 or higher treatment-emergent FN | 5
  Grade 3 or higher treatment-related treatment-emergent FN | 5

2. Primary Outcome: Complete Response (CR) Rate at EOT (Parts B and C)
Description: CR rate at EOT is defined as the percentage of participants with CR at EOT, according to the Lugano Classification Revised Staging System for malignant lymphoma (Cheson 2014) with the incorporation of Lymphoma Response to Immunomodulatory Therapy Criteria (LYRIC) (Cheson 2016), in participants with previously untreated cHL.
Time Frame: 7.8 months
Population: For Parts B and C, the full analysis set included all participants who enrolled and received any amount of the combination therapy in the study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part B | Part C
Number analyzed (Participants) | 57 | 154
Percentage of participants | 88 [76.3 to 94.9] | 92 [86.0 to 95.4]

3. Secondary Outcome: Number of Participants With Adverse Events of Clinical Interest (AECI) (Part A)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigational participant administered a medicinal product and which did not necessarily have a causal relationship with the treatment. Participants with peripheral neuropathy (PN) adverse events were summarized under AECI.
Time Frame: Approximately up to 7.5 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A
Number analyzed (Participants) | 40
Participants | 32

4. Secondary Outcome: Primary Refractory Disease Rate (Part A)
Description: The primary refractory disease rate is defined as the percentage of participants with less than complete response or relapse within 3 months of EOT, according to the Lugano Classification Revised Staging System for nodal non-Hodgkin and Hodgkin lymphomas
Time Frame: 10.2 months
Population: For Part A, the full analysis set includes all participants who received at least 1 dose of A+AVD (any of the study drugs in the regimen).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A
Number analyzed (Participants) | 40
percentage of participants | 10 [2.8 to 23.7]

5. Secondary Outcome: Complete Response Rate (Part A)
Description: The complete response rate is defined as the percentage of participants with CR at EOT according to the Lugano Classification Revised Staging System for nodal non-Hodgkin and Hodgkin lymphomas (Cheson 2014).
Time Frame: 7.2 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A
Number analyzed (Participants) | 40
percentage of participants | 80 [64.4 to 90.9]

6. Secondary Outcome: Physician-reported Progression Free Survival (PFS) (Part A)
Description: The physician-reported PFS rate at 2 years is estimated based on Kaplan-Meier methodology. The determination of antitumor activity will be based on response assessments made according to the Lugano Classification Revised Staging System for nodal non-Hodgkin and Hodgkin lymphomas (Cheson 2014).
Time Frame: 24 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A
Number analyzed (Participants) | 40
percentage of participants | 89.23 [73.76 to 95.82]

7. Secondary Outcome: Number of Participants With Subsequent Anticancer Therapy Utilization (Part A)
Description: Number of participants with subsequent anticancer therapy have been reported in this outcome measure.
Time Frame: 33.8 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part A
Number analyzed (Participants) | 40
Participants
  Participants with any subsequent therapy | 6
  Consolidative radiotherapy: Radiotherapy | 3
  Consolidative radiotherapy: Proton radiation | 1
  Immunotherapy: Nivolumab | 1
  Maintenance: Nivolumab | 1
  Maintenance radiotherapy: Radiation therapy | 1
  Systemic therapy for progressive disease: Bendamustine monotherapy | 1
  Systemic therapy for relapsed disease: Nivolumab | 1

8. Secondary Outcome: Actual Dose Intensity: Brentuximab Vedotin (Part A)
Time Frame: 6.5 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/kg/week
Arm/Group | Part A
Number analyzed (Participants) | 40
mg/kg/week | 0.5 (0.1)

9. Secondary Outcome: Actual Dose Intensity: Doxorubicin, Vinblastine, Dacarbazine (Part A)
Time Frame: 6.5 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/m2/week
Arm/Group | Part A
Number analyzed (Participants) | 40
mg/m2/week
  Doxorubicin | 11.8 (1.0)
  Vinblastine | 2.7 (0.4)
  Dacarbazine | 176.3 (15.2)

10. Secondary Outcome: Relative Dose Intensity (Part A)
Time Frame: 6.5 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of intended dose
Arm/Group | Part A
Number analyzed (Participants) | 40
percentage of intended dose
  Brentuximab vedotin | 91.0 (10.8)
  Doxorubicin | 94.2 (8.2)
  Vinblastine | 89.0 (13.6)
  Dacarbazine | 94.0 (8.1)

11. Secondary Outcome: Rate of Dose Reduction and Delays: Brentuximab Vedotin (Part A)
Time Frame: 6.5 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part A
Number analyzed (Participants) | 40
Participants
  Participants with any dose modification | 29
  Participants with any dose delay | 22
  Participants with any dose delay due to AE | 15
  Participants with any dose delay due to other reason | 14
  Participants with any dose reduction due to AE | 14

12. Secondary Outcome: Rate of Dose Reduction and Delays: Doxorubicin (Part A)
Time Frame: 6.5 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part A
Number analyzed (Participants) | 40
Participants
  Participants with any dose modification | 25
  Participants with any dose delay | 23
  Participants with any dose delay due to AE | 15
  Participants with any dose delay due to other reason | 15
  Participants with any dose reduction due to AE | 7

13. Secondary Outcome: Rate of Dose Reduction and Delays: Vinblastine (Part A)
Time Frame: 6.5 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part A
Number analyzed (Participants) | 40
Participants
  Participants with any dose modification | 27
  Participants with any dose delay | 22
  Participants with any dose delay due to AE | 15
  Participants with any dose delay due to other reason | 14
  Participants with any dose reduction due to AE | 12

14. Secondary Outcome: Rate of Dose Reduction and Delays: Dacarbazine (Part A)
Time Frame: 6.5 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part A
Number analyzed (Participants) | 40
Participants
  Participants with any dose modification | 25
  Participants with any dose delay | 22
  Participants with any dose delay due to AE | 15
  Participants with any dose delay due to other reason | 14
  Participants with any dose reduction due to AE | 6

15. Secondary Outcome: Incidence of Adverse Events (Parts B and C)
Time Frame: 8.9 months
Population: For Parts B and C, the full analysis set includes all participants who enrolled and received any amount of the combination therapy in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B | Part C
Number analyzed (Participants) | 57 | 154
Participants
  Any treatment-emergent adverse event (TEAE) | 57 | 153
  Treatment-related TEAE | 56 | 149
  Grade 3 or higher TEAE | 29 | 67
  Grade 3 or higher treatment-related TEAE | 19 | 52
  Any treatment-emergent serious adverse event (SAE) | 15 | 29
  Treatment-related treatment-emergent SAE | 8 | 19
  Participants who discontinued treatment due to TEAE | 4 | 4
  Participants who discontinued treatment due to treatment-related TEAE | 4 | 4
  TEAE leading to death | 0 | 0

16. Secondary Outcome: Incidence of Laboratory Abnormalities (Parts B and C)
Description: Laboratory values were graded according to the National Cancer Institute's (NCI) Common Terminology Criteria for Adverse Events (CTCAE version 4.03). As per NCI CTCAE version 4.03 grading, Grade 1 indicated mild or asymptomatic laboratory abnormalities, Grade 2 indicated moderate laboratory abnormalities, and Grade 3 indicated severe and 4 indicated life-threatening laboratory abnormalities.
Time Frame: 8.9 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part B | Part C
Number analyzed (Participants) | 57 | 154
Participants
  Hemoglobin high, Grade 1 | 0 | 4
  Hemoglobin high, Grade 2 | 0 | 0
  Hemoglobin high, Grade 3 | 0 | 0
  Hemoglobin high, Grade 4 | 0 | 0
  Hemoglobin low, Grade 1 | 37 | 96
  Hemoglobin low, Grade 2 | 10 | 6
  Hemoglobin low, Grade 3 | 1 | 1
  Hemoglobin low, Grade 4 | 0 | 0
  Leukocytes high, Grade 1 | 0 | 0
  Leukocytes high, Grade 2 | 0 | 0
  Leukocytes high, Grade 3 | 0 | 0
  Leukocytes high, Grade 4 | 0 | 0
  Leukocytes low, Grade 1 | 19 | 41
  Leukocytes low, Grade 2 | 12 | 24
  Leukocytes low, Grade 3 | 0 | 2
  Leukocytes low, Grade 4 | 0 | 0
  Lymphocytes high, Grade 1 | 0 | 0
  Lymphocytes high, Grade 2 | 1 | 3
  Lymphocytes high, Grade 3 | 0 | 0
  Lymphocytes high, Grade 4 | 0 | 0
  Lymphocytes low, Grade 1 | 11 | 31
  Lymphocytes low, Grade 2 | 17 | 22
  Lymphocytes low, Grade 3 | 7 | 9
  Lymphocytes low, Grade 4 | 1 | 0
  Neutrophils low, Grade 1 | 4 | 12
  Neutrophils low, Grade 2 | 14 | 38
  Neutrophils low, Grade 3 | 4 | 11
  Neutrophils low, Grade 4 | 2 | 3
  Platelets low, Grade 1 | 6 | 22
  Platelets low, Grade 2 | 1 | 1
  Platelets low, Grade 3 | 0 | 0
  Platelets low, Grade 4 | 0 | 0
  Alanine aminotransferase high, Grade 1 | 26 | 71
  Alanine aminotransferase high, Grade 2 | 3 | 16
  Alanine aminotransferase high, Grade 3 | 4 | 10
  Alanine aminotransferase high, Grade 4 | 0 | 0
  Albumin low, Grade 1 | 11 | 22
  Albumin low, Grade 2 | 3 | 6
  Albumin low, Grade 3 | 0 | 0
  Albumin low, Grade 4 | 0 | 0
  Alkaline phosphatase high, Grade 1 | 30 | 51
  Alkaline phosphatase high, Grade 2 | 2 | 1
  Alkaline phosphatase high, Grade 3 | 0 | 0
  Alkaline phosphatase high, Grade 4 | 0 | 0
  Amylase high, Grade 1 | 3 | 15
  Amylase high, Grade 2 | 2 | 6
  Amylase high, Grade 3 | 0 | 6
  Amylase high, Grade 4 | 0 | 0
  Aspartate aminotransferase high, Grade 1 | 27 | 75
  Aspartate aminotransferase high, Grade 2 | 1 | 7
  Aspartate aminotransferase high, Grade 3 | 2 | 1
  Aspartate aminotransferase high, Grade 4 | 0 | 0
  Calcium corrected for albumin high, Grade 1 | 12 | 18
  Calcium corrected for albumin high, Grade 2 | 0 | 0
  Calcium corrected for albumin high, Grade 3 | 0 | 0
  Calcium corrected for albumin high, Grade 4 | 0 | 0
  Calcium corrected for albumin low, Grade 1 | 7 | 5
  Calcium corrected for albumin low, Grade 2 | 0 | 1
  Calcium corrected for albumin low, Grade 3 | 0 | 0
  Calcium corrected for albumin low, Grade 4 | 0 | 0
  Ionized calcium high, Grade 1 | 0 | 0
  Ionized calcium high, Grade 2 | 0 | 0
  Ionized calcium high, Grade 3 | 0 | 0
  Ionized calcium high, Grade 4 | 0 | 0
  Ionized calcium low, Grade 1 | 0 | 0
  Ionized calcium low, Grade 2 | 0 | 0
  Ionized calcium low, Grade 3 | 0 | 0
  Ionized calcium low, Grade 4 | 0 | 0
  Creatinine high, Grade 1 | 47 | 127
  Creatinine high, Grade 2 | 5 | 11
  Creatinine high, Grade 3 | 1 | 0
  Creatinine high, Grade 4 | 0 | 0
  Estimated glomerular filtration rate low, Grade 1 | 1 | 8
  Estimated glomerular filtration rate low, Grade 2 | 4 | 10
  Estimated glomerular filtration rate low, Grade 3 | 0 | 0
  Estimated glomerular filtration rate low, Grade 4 | 0 | 0
  Glucose high, Grade 1 | 45 | 69
  Glucose high, Grade 2 | 5 | 9
  Glucose high, Grade 3 | 1 | 13
  Glucose high, Grade 4 | 1 | 0
  Glucose low, Grade 1 | 12 | 18
  Glucose low, Grade 2 | 1 | 0
  Glucose low, Grade 3 | 0 | 0
  Glucose low, Grade 4 | 0 | 0
  Lipase high, Grade 1 | 9 | 13
  Lipase high, Grade 2 | 1 | 6
  Lipase high, Grade 3 | 5 | 6
  Lipase high, Grade 4 | 0 | 3
  Phosphate low, Grade 1 | 1 | 3
  Phosphate low, Grade 2 | 7 | 9
  Phosphate low, Grade 3 | 2 | 4
  Phosphate low, Grade 4 | 0 | 0
  Potassium high, Grade 1 | 3 | 7
  Potassium high, Grade 2 | 0 | 1
  Potassium high, Grade 3 | 0 | 0
  Potassium high, Grade 4 | 0 | 0
  Potassium low, Grade 1 | 9 | 19
  Potassium low, Grade 2 | 0 | 0
  Potassium low, Grade 3 | 2 | 0
  Potassium low, Grade 4 | 1 | 0
  Sodium high, Grade 1 | 2 | 3
  Sodium high, Grade 2 | 0 | 0
  Sodium high, Grade 3 | 0 | 1
  Sodium high, Grade 4 | 0 | 0
  Sodium low, Grade 1 | 11 | 25
  Sodium low, Grade 2 | 0 | 0
  Sodium low, Grade 3 | 2 | 2
  Sodium low, Grade 4 | 0 | 0
  Total bilirubin high, Grade 1 | 1 | 8
  Total bilirubin high, Grade 2 | 2 | 0
  Total bilirubin high, Grade 3 | 0 | 0
  Total bilirubin high, Grade 4 | 0 | 0
  Urate high, Grade 1 | 0 | 0
  Urate high, Grade 2 | 0 | 0
  Urate high, Grade 3 | 10 | 28
  Urate high, Grade 4 | 0 | 1

17. Secondary Outcome: Overall Response Rate (ORR) at EOT (Parts B and C)
Description: ORR is defined as the percentage of participants with CR or partial response (PR) at EOT according to the Lugano Classification Revised Staging System for malignant lymphoma (Cheson 2014) with the incorporation of LYRIC (Cheson 2016) in participants with previously untreated cHL.
Time Frame: Up to 7.8 months
Population: For Parts B and C, the full analysis set included all participants who were enrolled and received any amount of the combination therapy in the study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part B | Part C
Number analyzed (Participants) | 57 | 154
Percentage of participants | 93 [83.0 to 98.1] | 96 [91.7 to 98.6]

18. Secondary Outcome: Duration of Response (DOR) at End of Study (Parts B and C)
Description: DOR was defined as the time from the first documentation of objective tumor response (CR or PR) to the first documentation of tumor progression per the Lugano Classification Revised Staging System for malignant lymphoma (Cheson 2014) with the incorporation of LYRIC (Cheson 2016) or death, whichever came first. Duration of response was only calculated for the subgroup of participants achieving a CR or PR. Participants without progression or death were censored on the date of the last radiological assessment of measured lesions. Kaplan-Meier method was used.
Time Frame: Up to 51.1 months
Population: For Parts B and C, the full analysis set includes all participants who were enrolled and received any amount of the combination therapy in the study. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part B | Part C
Number analyzed (Participants) | 56 | 154
Months | NA [NA to NA] — Median and 95% CI were not estimable due to insufficient number of participants with event. | NA [NA to NA] — Median and 95% CI were not estimable due to insufficient number of participants with event.

19. Secondary Outcome: Duration of Complete Response (DOCR) (Parts B and C)
Description: DOCR was defined as the time from start of the first documentation of CR to the first documentation of tumor progression (per the Lugano Classification Revised Staging System for malignant lymphoma (Cheson 2014) with the incorporation of LYRIC (Cheson 2016) or death, whichever came first. DOCR was calculated for the subgroup of participants achieving CR. Participants without progression or death were censored on the date of the last radiological assessment of measured lesions. Kaplan-Meier method was used.
Time Frame: Up to 51.1 months
Population: as for outcome 18
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part B | Part C
Number analyzed (Participants) | 56 | 154
Months | NA [NA to NA] — Median and 95% CI were not estimable due to insufficient number of participants with event. | NA [NA to NA] — Median and 95% CI were not estimable due to insufficient number of participants with event.

20. Secondary Outcome: Event Free Survival (EFS) Rate (Parts B and C)
Description: EFS was defined as the time from the start of study treatment to the first documentation of objective tumor progression, death due to any cause, or receipt of subsequent anticancer therapy to treat residual or progressive disease, whichever occurred first. The determination of antitumor activity will be based on objective response assessments made according to Lugano Classification Revised Staging System for malignant lymphoma (Cheson 2014) with the incorporation of LYRIC (Cheson 2016). Participants without progression or death were censored on the date of the last radiological assessment of measured lesions. EFS rate was percentage of participants with EFS.
Time Frame: Months 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39 and 42
Population: For Parts B and C, the full analysis set includes all participants who were enrolled and received any amount of the combination therapy in the study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part B | Part C
Number analyzed (Participants) | 57 | 154
Percentage of participants
  Month 3 | 98.25 [88.19 to 99.75] | 100 [100 to 100]
  Month 6 | 98.25 [88.19 to 99.75] | 98.66 [94.74 to 99.66]
  Month 9 | 94.67 [84.39 to 98.25] | 98.66 [94.74 to 99.66]
  Month 12 | 92.89 [82.15 to 97.27] | 98.66 [94.74 to 99.66]
  Month 15 | 91.03 [79.77 to 96.17] | 97.95 [93.79 to 99.34]
  Month 18 | 91.03 [79.77 to 96.17] | 96.46 [91.70 to 98.51]
  Month 21 | 86.89 [74.38 to 93.55] | 96.46 [91.70 to 98.51]
  Month 24 | 86.89 [74.38 to 93.55] | 95.62 [90.49 to 98.02]
  Month 27 | 86.89 [74.38 to 93.55] | 94.72 [89.19 to 97.46]
  Month 30 | 86.89 [74.38 to 93.55] | 94.72 [89.19 to 97.46]
  Month 33 | 84.54 [71.29 to 92.01] | 94.72 [89.19 to 97.46]
  Month 36 | 84.54 [71.29 to 92.01] | 94.72 [89.19 to 97.46]
  Month 39 | 84.54 [71.29 to 92.01] | 94.72 [89.19 to 97.46]
  Month 42: number analyzed (Participants) | 57 | 0
  Month 42 | 84.54 [71.29 to 92.01] |

21. Secondary Outcome: PFS Rate (Parts B and C)
Description: PFS was defined as the time from start of study treatment to first documentation of objective tumor progression or death. The determination of antitumor activity will be based on objective response assessments made according to Lugano Classification Revised Staging System for malignant lymphoma (Cheson 2014) with the incorporation of LYRIC (Cheson 2016). Participants without progression or death were censored on the date of the last radiological assessment of measured lesions. Kaplan-Meier method was used.
Time Frame: At months 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39 and 42 from the start of study treatment
Population: as for outcome 20
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part B | Part C
Number analyzed (Participants) | 57 | 154
Percentage of participants
  Month 3 | 100 [100 to 100] | 100 [100 to 100]
  Month 6 | 100 [100 to 100] | 100 [100 to 100]
  Month 9 | 96.36 [86.23 to 99.08] | 100 [100 to 100]
  Month 12 | 94.55 [84.04 to 98.21] | 100 [100 to 100]
  Month 15 | 92.65 [81.59 to 97.18] | 99.29 [95.04 to 99.90]
  Month 18 | 92.65 [81.59 to 97.18] | 97.77 [93.26 to 99.28]
  Month 21 | 88.44 [76.00 to 94.65] | 97.77 [93.26 to 99.28]
  Month 24 | 88.44 [76.00 to 94.65] | 96.92 [91.99 to 98.84]
  Month 27 | 88.44 [76.00 to 94.65] | 96.01 [90.64 to 98.33]
  Month 30 | 88.44 [76.00 to 94.65] | 96.01 [90.64 to 98.33]
  Month 33 | 86.05 [72.80 to 93.14] | 96.01 [90.64 to 98.33]
  Month 36 | 86.05 [72.80 to 93.14] | 96.01 [90.64 to 98.33]
  Month 39 | 86.05 [72.80 to 93.14] | 96.01 [90.64 to 98.33]
  Month 42: number analyzed (Participants) | 57 | 0
  Month 42 | 86.05 [72.80 to 93.14] |

22. Secondary Outcome: Overall Survival (OS) Rate (Parts B and C)
Description: OS was defined as the time from start of study treatment to date of death due to any cause. In the absence of confirmation of death, survival time was censored at the last date the participant was known to be alive. Kaplan-Meier method was used.
Time Frame: At months 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39 and 42 from the start of study treatment
Population: as for outcome 20
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part B | Part C
Number analyzed (Participants) | 57 | 154
Percentage of participants
  Month 3 | 100 [100 to 100] | 100 [100 to 100]
  Month 6 | 100 [100 to 100] | 100 [100 to 100]
  Month 9 | 100 [100 to 100] | 100 [100 to 100]
  Month 12 | 98.25 [88.19 to 99.75] | 100 [100 to 100]
  Month 15 | 98.25 [88.19 to 99.75] | 100 [100 to 100]
  Month 18 | 98.25 [88.19 to 99.75] | 100 [100 to 100]
  Month 21 | 98.25 [88.19 to 99.75] | 100 [100 to 100]
  Month 24 | 98.25 [88.19 to 99.75] | 100 [100 to 100]
  Month 27 | 98.25 [88.19 to 99.75] | 100 [100 to 100]
  Month 30 | 98.25 [88.19 to 99.75] | 100 [100 to 100]
  Month 33 | 98.25 [88.19 to 99.75] | 98.73 [91.35 to 99.82]
  Month 36 | 98.25 [88.19 to 99.75] | 98.73 [91.35 to 99.82]
  Month 39 | 98.25 [88.19 to 99.75] | 98.73 [91.35 to 99.82]
  Month 42 | 98.25 [88.19 to 99.75] | 98.73 [91.35 to 99.82]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: Up to 54.5 Months, Serious Adverse Events, and Non-Serious Adverse Events were followed for up to 8.9 months.
Description: The population for all-cause mortality and adverse events includes participants who received at least one dose of study drug.
Arm/Group | Part A | Part B | Part C
All-Cause Mortality (participants affected / at risk) | 2/40 | 1/57 | 1/154
Serious Adverse Events (participants affected / at risk) | 19/40 | 15/57 | 29/154
Other Adverse Events (participants affected / at risk) | 40/40 | 57/57 | 153/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A (N=40) | Part B (N=57) | Part C (N=154)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 3 (4) | 6 (7)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Autoimmune disorder (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Meningitis aseptic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 4 (5) | 0 (0) | 2 (2)
Pneumonia fungal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash morbilliform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A (N=40) | Part B (N=57) | Part C (N=154)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 6 (6) | 8 (10)
Anaemia folate deficiency (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (5)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (9) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (7) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (6) | 6 (10) | 19 (22)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 2 (2)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 8 (9)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 2 (2) | 6 (6)
Tachycardia (Cardiac disorders) | 4 (4) | 1 (1) | 3 (3)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
External ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 7 (8)
Hypothyroidism (Endocrine disorders) | 0 (0) | 5 (5) | 10 (10)
Immune-mediated thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Thyroid mass (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2)
Chalazion (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 2 (2) | 5 (5)
Epiretinal membrane (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 2 (2) | 3 (3) | 2 (2)
Photophobia (Eye disorders) | 1 (3) | 1 (1) | 0 (0)
Photopsia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 4 (6) | 6 (6) | 7 (7)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Vitreous detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Xerophthalmia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 2 (2) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 10 (11) | 6 (11) | 15 (17)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 18 (22) | 22 (24) | 69 (86)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 13 (17) | 26 (33) | 38 (49)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 2 (2) | 9 (9)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 6 (6) | 15 (16)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (5) | 5 (5) | 17 (17)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Glossitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (2) | 2 (2)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 4 (4) | 4 (4)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lip oedema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lip pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 28 (31) | 40 (58) | 105 (135)
Noninfective sialoadenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophageal dilatation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oral dysaesthesia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 5 (5)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 9 (11) | 9 (9) | 23 (27)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 9 (12) | 16 (17) | 25 (33)
Asthenia (General disorders) | 0 (0) | 0 (0) | 2 (2)
Axillary pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Catheter site bruise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Catheter site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Catheter site inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 6 (6)
Catheter site rash (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 6 (7)
Chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
Chills (General disorders) | 3 (3) | 5 (6) | 6 (6)
Face oedema (General disorders) | 0 (0) | 0 (0) | 2 (2)
Facial pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 15 (16) | 29 (36) | 74 (83)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 6 (6)
Infusion site pain (General disorders) | 0 (0) | 0 (0) | 2 (3)
Infusion site pruritus (General disorders) | 1 (1) | 0 (0) | 0 (0)
Infusion site rash (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 2 (3)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 1 (1)
Malaise (General disorders) | 2 (2) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (2) | 3 (4) | 8 (8)
Oedema peripheral (General disorders) | 5 (5) | 3 (4) | 6 (7)
Pain (General disorders) | 2 (2) | 4 (4) | 6 (6)
Peripheral swelling (General disorders) | 0 (0) | 2 (2) | 0 (0)
Puncture site swelling (General disorders) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 8 (8) | 6 (9) | 21 (28)
Swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Swelling face (General disorders) | 0 (0) | 1 (1) | 1 (1)
Temperature intolerance (General disorders) | 0 (0) | 1 (1) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (4)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (3)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 1 (1) | 4 (6)
Contrast media allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 3 (3) | 24 (27)
Candida infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Epstein-Barr virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Fungal foot infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (3)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 2 (3) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infected bite (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Klebsiella infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nail bed infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Omphalitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 3 (3) | 4 (4)
Oral herpes (Infections and infestations) | 0 (0) | 2 (3) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Penile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Peripheral nerve infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pilonidal disease (Infections and infestations) | 1 (2) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 4 (4)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Prostate infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Systemic candida (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 3 (3) | 11 (13)
Urinary tract infection (Infections and infestations) | 0 (0) | 6 (8) | 5 (6)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 4 (4) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 14 (19)
Injection related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 2 (2)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (5) | 9 (11) | 33 (50)
Amylase increased (Investigations) | 0 (0) | 2 (3) | 11 (16)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 7 (8) | 27 (36)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 2 (3) | 4 (4)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 2 (7) | 3 (3)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 3 (3)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Fibrin D dimer increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (4)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Heart rate irregular (Investigations) | 0 (0) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (2) | 6 (7)
Liver function test increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (1) | 3 (5)
Neutrophil count decreased (Investigations) | 5 (5) | 5 (7) | 5 (9)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 6 (6) | 5 (5) | 10 (10)
Weight increased (Investigations) | 1 (1) | 6 (7) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 2 (4)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 11 (12) | 9 (10) | 22 (29)
Dehydration (Metabolism and nutrition disorders) | 5 (25) | 4 (5) | 5 (5)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Food aversion (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (5) | 3 (3)
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 6 (8)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (3) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 9 (13) | 5 (6)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (4) | 2 (3) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 7 (9) | 16 (19)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 6 (6) | 16 (16)
Bone pain (Musculoskeletal and connective tissue disorders) | 12 (14) | 10 (10) | 10 (11)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 4 (7)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 4 (4)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (8) | 8 (12) | 12 (12)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 4 (4)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (8) | 4 (4) | 9 (11)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (4)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour thrombosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 2 (2) | 1 (1) | 4 (4)
Dizziness (Nervous system disorders) | 10 (12) | 6 (7) | 16 (18)
Dysaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 9 (9) | 5 (5) | 13 (14)
Headache (Nervous system disorders) | 13 (14) | 15 (20) | 36 (46)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 3 (3) | 1 (2) | 1 (1)
Intensive care unit acquired weakness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Neuropathy peripheral (Nervous system disorders) | 2 (3) | 0 (0) | 2 (2)
Neurotoxicity (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 2 (2) | 2 (2) | 7 (9)
Parosmia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 4 (4) | 1 (1) | 2 (2)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 25 (34) | 26 (34) | 72 (79)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Taste disorder (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2) | 8 (9) | 16 (16)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 2 (2) | 2 (2) | 4 (4)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Drug abuse (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 11 (11) | 6 (6) | 21 (21)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Restlessness (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Immune-mediated nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Lower urinary tract symptoms (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urine abnormality (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Menstrual disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 3 (3) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Premature menopause (Reproductive system and breast disorders) | 0 (0) | 4 (4) | 2 (2)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 1 (1)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (7) | 18 (19)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 10 (11) | 26 (29)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 8 (8)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 6 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 10 (10)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 2 (2) | 13 (14)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 5 (5)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 3 (3)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper airway resistance syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 5 (6) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 12 (12) | 21 (21) | 34 (34)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (5) | 3 (5)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 5 (5)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 3 (3)
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 6 (7)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 4 (4)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 5 (5)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Penile ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5) | 13 (13)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 4 (6) | 13 (15)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (8) | 11 (12) | 20 (28)
Rash morbilliform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Umbilical erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Urticaria chronic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Catheter placement (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Cyst drainage (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Vocal cord polypectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Wisdom teeth removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Cyanosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 2 (2) | 2 (2)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 2 (4) | 5 (5)
Hot flush (Vascular disorders) | 3 (3) | 7 (7) | 11 (12)
Hypertension (Vascular disorders) | 1 (1) | 4 (4) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 2 (3) | 4 (4)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 3 (3)
Superficial vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Withdrawal hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-07-31): https://cdn.clinicaltrials.gov/large-docs/23/NCT03646123/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-27): https://cdn.clinicaltrials.gov/large-docs/23/NCT03646123/SAP_001.pdf